CLINICAL TRIAL: NCT06691620
Title: Effects of Different Nasal Irrigation Methods on Pain Level, Crying and Procedure Times, and Physiologic Parameters in Nasal Congestion in Infants: a Randomized Controlled Trial
Brief Title: Effects of Different Nasal Irrigation Methods on Pain Level, Crying and Procedure Times in Nasal Congestion in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-01-22
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Nasal Congestion; Nursing
Keywords: Infant; nasal congestion; nasal irrigation; nasopharyngeal aspiration; nursing
MeSH Terms: conditions — Nasal Obstruction | interventions — Nasal Lavage; Sodium Chloride; Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Participants were assigned to the groups using the block randomization method. Age (6-12 and 13-24 months) and sex (male and female) were used as variables for randomization. Blocks were repeated eight times in each group to achieve the calculated sample size, and 32 participants were included in each group. An online tool was used to generate the randomization list with 2 × 2 × 8 blocks (Sealed Envelope Ltd., 2022).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Using the block randomization technique, participants were divided into four groups. A web-based randomization list generation tool was used to assign participants to groups. Control and intervention groups were coded as A, B, C and D using the sealed envelope method. Randomization information was withheld from the researcher involved in data collection until data was collected. The researcher determines which group each baby is in. The researcher found out during the painful procedure. (investigator blinding). Within the scope of the research, parents knew which group the baby was in. However, due to the nature of the sample group, the babies were blind. To avoid statistical bias, study groups were coded as A, B, C and D; statistical blinding was performed (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention 1 Group (Experimental): The group received a nasal irrigation procedure with isotonic saline.
  Interventions: Procedure: Nasal irrigation with isotonic saline
- Intervention 2 Group (Experimental): The group received a nasal irrigation procedure with hypertonic saline.
  Interventions: Procedure: Nasal irrigation with hypertonic saline
- Intervention 3 Group (Experimental): The group received a nasal irrigation procedure with isotonic saline and nontraumatic nasopharyngeal aspiration.
  Interventions: Procedure: Nasal irrigation with isotonic saline; Procedure: Nontraumatic nasopharyngeal aspiration
- Intervention 4 Group (Experimental): The group received a nasal irrigation procedure with hypertonic saline and nontraumatic nasopharyngeal aspiration.
  Interventions: Procedure: Nasal irrigation with hypertonic saline; Procedure: Nontraumatic nasopharyngeal aspiration

INTERVENTIONS:
Procedure: Nasal irrigation with isotonic saline — Infants were placed on the examination stretcher in the right or left lateral position. Then, 10 mL of isotonic saline solution was administered over 5 s into the upper nasal cavity of the infant. The secretion and irrigation solution from the lower nasal cavity were cleaned using gauze. The infant was placed on the other side, and the same procedure was repeated for the other nasal cavity. The infant was then placed in the prone position, and the tapotement technique was applied. The infant's mouth and nose were cleaned with gauze, completing the procedure.
  Arms: Intervention 1 Group; Intervention 3 Group
Procedure: Nasal irrigation with hypertonic saline — Infants were placed on the examination stretcher in the right or left lateral position. Then, 10 mL of hypertonic saline solution was administered over 5 s into the upper nasal cavity of the infant. The secretion and irrigation solution from the lower nasal cavity were cleaned using gauze. The infant was placed on the other side, and the same procedure was repeated for the other nasal cavity. The infant was then placed in the prone position, and the tapotement technique was applied. The infant's mouth and nose were cleaned with gauze, completing the procedure.
  Arms: Intervention 2 Group; Intervention 4 Group
Procedure: Nontraumatic nasopharyngeal aspiration — After nasal irrigation, the secretions and saline solution from the underlying nasal cavity were nontraumatically aspirated from the entrance of the nasal cavity after the irrigation. The infant was positioned on the other side, and the same procedure was repeated for the other nasal cavity. The infant was then placed in the prone position, and the tapotement technique was applied. The infant's mouth and nose were cleaned with gauze, completing the procedure.
  Arms: Intervention 3 Group; Intervention 4 Group

SUMMARY:
This study aimed to evaluate the effects of different nasal irrigation (NI) methods for relieving nasal obstruction on pain, crying and procedure times, and physiologic parameters in infants with acute upper respiratory tract infection.

DETAILED DESCRIPTION:
Acute upper respiratory tract infections (URTIs) are the leading cause of acute disease incidence worldwide. Nasal saline irrigation (NSI) is a recommended approach to relieve nasal symptoms and maintain upper airway patency in children, offering a safe, inexpensive, and well-tolerated symptomatic treatment for children with URTIs. Nasal irrigation (NI) relieves URTI symptoms by clearing mucus, reducing congestion, and improving breathing. NI techniques and irrigation solutions used to relieve nasal obstruction in infants are effective in providing procedural comfort. Considering the effectiveness of NI in relieving nasal congestion, which negatively influences the quality of life of children, filling the gap in the literature on NSI is crucial. This study was conducted to determine the effects of various NI methods (NI/NI + nontraumatic nasopharyngeal aspiration) using different irrigation solutions on pain, crying and procedure times, and physiologic parameters in infants with URTIs aged 6 months to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* infants aged between 6 months and 24 months, born at term, and recommended NSI for nasal cleansing by the physician due to a diagnosis of URTI.

Exclusion Criteria:

* infants with chronic diseases, nasal congestion due to reasons other than URTI, congenital anomalies related to the respiratory system, allergic rhinitis, unconsciousness, use of analgesics, antibiotics, and corticosteroids before admission to the hospital, and developmental retardation.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Procedural pain score- FLACC Pain Scale | 1 minute before the heel lance procedure, at the end of the procedure
  The Face, Legs, Activity, Cry, and Consolability (FLACC) scale consists of five categories (face, legs, activity, crying, and consolability), and each category is scored between 0 and 2 depending on the pain or distress behaviors observed. The total score ranges from 0 to 10, with 0 indicating no pain or distress and 10 indicating extreme pain or distress. The FLACC scale was developed to assess pain in children aged 2 months to 7 years and is one of the widely recommended scales for assessing pain and distress among pediatric patients.
Crying time | Through painful procedure completion, an average of 5 minutes
  The crying time was the duration of infants' crying from the start of the NI procedure to 5 min after the procedure.
Procedure time | Through painful procedure completion, an average of 2 minutes.
  The procedure started with positioning the infant to apply NI in the first nasal cavity and ended with the completion of NI in the second nasal cavity

SECONDARY OUTCOMES:
SpO2 | 1 minute before the procedure, at the end of the procedure, and 5 min after the procedure.
  In this study, SpO2 values of infants were measured 3 times.
Heart rate /minute | 1 minute before the procedure, at the end of the procedure, and and 5 min after the procedure.
  In this study, heart rate /minute values of infants were measured 3 times.
Respiratory rate/ minute | 1 minute before the procedure, at the end of the procedure, and 5 min after the procedure.
  In this study, Respiratory rate/ minute values of infants were measured 3 times.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, Professor, Study Director — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Kadıköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: September through December of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Avşar Gök, N. & Bozkurt, G. (2023). Effects of two different nasal irrigation techniques on physiological parameters and crying duration in relieving nasal congestion in infants. Authorea, in press
- [Background] Koksal T, Cizmeci MN, Bozkaya D, Kanburoglu MK, Sahin S, Tas T, Yuksel CN, Tatli MM. Comparison between the use of saline and seawater for nasal obstruction in children under 2 years of age with acute upper respiratory infection. Turk J Med Sci. 2016 Jun 23;46(4):1004-13. doi: 10.3906/sag-1507-18. PMID 27513397
- [Background] Cabaillot A, Vorilhon P, Roca M, Boussageon R, Eschalier B, Pereirad B. Saline nasal irrigation for acute upper respiratory tract infections in infants and children: A systematic review and meta-analysis. Paediatr Respir Rev. 2020 Nov;36:151-158. doi: 10.1016/j.prrv.2019.11.003. Epub 2020 Feb 21. PMID 32312677